CLINICAL TRIAL: NCT04645394
Title: Bioavailability of Anthocyanins From Aronia Extract
Brief Title: Bioavailability of Anthocyanins From Aronia Extract in Healthy Men - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1-10-72-57-20
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2020-11

CONDITIONS: Bioavailability
Keywords: bioavailability; Aronia melanocarpa; polyphenols; anthocyanins; healthy; men; uptake
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: Acute 4-arm crossover intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): The participants are receiving 1 dose of each in the stated order.
  Interventions: Dietary Supplement: Aronia melanocarpa; Dietary Supplement: Fermented Aronia Melanocarpa high dose; Dietary Supplement: Fermented Aronia Melanocarpa low dose; Dietary Supplement: Placebo
- Fermented aronia high dose (Active Comparator): The participants are receiving 1 dose of each in the stated order.
  Interventions: Dietary Supplement: Aronia melanocarpa; Dietary Supplement: Fermented Aronia Melanocarpa high dose; Dietary Supplement: Fermented Aronia Melanocarpa low dose; Dietary Supplement: Placebo
- Fermented aronia low dose (Active Comparator): The participants are receiving 1 dose of each in the stated order.
  Interventions: Dietary Supplement: Aronia melanocarpa; Dietary Supplement: Fermented Aronia Melanocarpa high dose; Dietary Supplement: Fermented Aronia Melanocarpa low dose; Dietary Supplement: Placebo
- Aronia (Active Comparator): The participants are receiving 1 dose of each in the stated order.
  Interventions: Dietary Supplement: Aronia melanocarpa; Dietary Supplement: Fermented Aronia Melanocarpa high dose; Dietary Supplement: Fermented Aronia Melanocarpa low dose; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Aronia melanocarpa — Administered once (acute study)
  Other Names: Chokeberry
Dietary Supplement: Fermented Aronia Melanocarpa high dose — Administered once (acute study)
  Other Names: Chokeberry
Dietary Supplement: Fermented Aronia Melanocarpa low dose — Administered once (acute study)
  Other Names: Chokeberry
Dietary Supplement: Placebo — Administered once (acute study)

SUMMARY:
In a quadruple cross-over design, 8 healthy men will receive 3 different formulations of Aronia extract as well as placebo (placebo, aronia, and fermented aronia in 1/6 and 1/1 concentration). The intervention will be given on four separate days at least three days apart. Before consumption, 2 fasting blood samples will be taken. Blood will also be sampled at 60, 120, 240, and 360 minutes post consumption. The blood samples will be analyzed for polyphenolic content with a special focus on anthocyanins.

DETAILED DESCRIPTION:
Methods for possible intervention The trial will be executed in accordance with the guidelines of the declaration of Helsinki and will be approved by The Danish Ethical Committee (1-10-72-57-20). The study is designed as a randomized acute-crossover study repeated on 4 separate days. All participants will be screened, and written consent must be obtained before the initiation of the study. Prior to the first intervention day, participants will be randomized to the order of the intervention; placebo, 1/6 mg or 1/1 fermented aronia extract or non-fermented aronia extract. In order to prevent any cross contamination between intervention days, no less than 3 washout days must pass between intervention days. Participants must be fasting for at least 8 hours with only water allowed.

Participants Participants will be recruited by advertisements as well as social media. Potential candidates will afterwards be referred to the head of the study who will orally explain the study. Provided interest from candidate, a written consent must be obtained. Participants will have the right to end their participation at any given point.

Intervention day and blood collections On intervention days, participants arrive fasting (water allowed since midnight). The intervention will be randomized as to which of the four interventions the participants are going to consume on the day. All participants will consume each intervention of either placebo, 1/6 or 1/1 dose fermented aronia extract or 1/1 dose from non-fermented aronia extract. 15 mins prior to consuming the intervention, a blood sample will be collected. Another sample will be collected at time 0 h, after which time the aronia extract along with 200 mL water must be consumed. Then, at time 60, 120, 240 and 360 min, blood must be collected also. At least 3 washout days must pass between intervention to ensure no cross contamination.

Biochemical analysis Following a successful collection of 6 blood samples over the course of 360 mins on intervention day, the blood from each participant will be stored at -80°C until analysis. The blood samples will be coded in an anonymous way to ensure that blood sample cannot be connected to participant to ensure anonymity. The analysis can be carried out by means of high-pressure liquid chromatography (HPLC) or an equivalent method. The blood samples must be evaluated for their possible anthocyanin content as well as their phenolic compound content.

Statistical analysis Primary outcome is area under the curve (total and incremental) for the response curves of anthocyanins.

To determine differences between groups, ANOVA test will be carried out. Data are considered significant if p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* man between ≥20 ≤75 years of age

Exclusion Criteria:

* Daily usage of medicine, alcohol- or substance abuse
* BMI ≥30

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
area under the curve for anthocyanin blood concentration | -15, 0, 60, 120, 240, 360 minutes
  Blood is sampled before (-15, 0) and after (60, 120, 240, 360) consumption
incremental area under the curve for anthocyanin blood concentration | -15, 0, 60, 120, 240, 360 minutes
  Blood is sampled before (-15, 0) and after (60, 120, 240, 360) consumption

SECONDARY OUTCOMES:
Concentration of polyphenols in the blood | -15, 0, 60, 120, 240, 360 minutes
  Blood is sampled before (-15, 0) and after (60, 120, 240, 360) consumption
Antioxidant activity in the blood | -15, 0, 60, 120, 240, 360 minutes
  Blood is sampled before (-15, 0) and after (60, 120, 240, 360) consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Danmark, Denmark